CLINICAL TRIAL: NCT03431740
Title: Fractional Exhaled NO, Extended NO Analysis and NO/CO Diffusing Capacity in Patients Receiving Thoracic Radiation Therapy: a Single Centre Study
Brief Title: FENO, Extended NO Analysis and NO/CO Diffusing Capacity in Thoracic Radiation Therapy
Status: Terminated | Type: Observational
Why Stopped: Insufficient recruitment
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-01374
Record Dates: First submitted 2018-01-18; First posted 2018-02-13 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2021-04

CONDITIONS: Radiotherapy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators aim to investigate the impact of thoracic radiation therapy on diffusion capacity of the lung (primary endpoint: diffusion capacity for nitric oxide, DLNO) and on exhaled nitric oxide.

ELIGIBILITY:
Inclusion Criteria:

* planned but not already commenced radiation therapy (RT) of the chest, with or without pre-RT surgery.
* signed informed consent of the participant

Exclusion Criteria:

* thoracic RT in the past
* treatment with immune checkpoint inhibitors
* unstable condition affecting participation in the measurements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists in patients with planned but not already commenced radiation therapy of the chest. Recruitment will be performed at the Radiation Oncology Clinic at University Hospital of Zurich.
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2018-02-15 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Change in diffusing capacity for nitric oxide (DLNO) | Before start of radiation therapy (RT), at the day of end of RT, 6 weeks and 12 months after end of RT

SECONDARY OUTCOMES:
Diffusing capacity for carbon monoxide (DLCO) | Before start of radiation therapy (RT), at the day of end of RT, 6 weeks and 12 months after end of RT
  The course over time will be described.
Transfer Coefficient for nitric oxide (DLNO/VA) | Before start of radiation therapy (RT), at the day of end of RT, 6 weeks and 12 months after end of RT
  The course over time will be described.
Transfer Coefficient for carbon monoxide (DLCO/VA) | Before start of radiation therapy (RT), at the day of end of RT, 6 weeks and 12 months after end of RT
  The course over time will be described.
Ratio of DLNO and DLCO | Before start of radiation therapy (RT), at the day of end of RT, 6 weeks and 12 months after end of RT
  The course over time will be described.
Alveolar-capillary membrane-diffusing capacity for carbon monoxide (DMCO) | Before start of radiation therapy (RT), at the day of end of RT, 6 weeks and 12 months after end of RT
  The course over time will be described.
Pulmonary capillary blood volume (Vc) | Before start of radiation therapy (RT), at the day of end of RT, 6 weeks and 12 months after end of RT
  This variable is a calculated variable. The course over time will be described.
Alveolar Volume (VA) | Before start of radiation therapy (RT), at the day of end of RT, 6 weeks and 12 months after end of RT
  This variable is a calculated variable. The course over time will be described.
Fractional concentration of exhaled nitric oxide at a flow rate of 50mL/s (FENO50) | Before start of radiation therapy (RT), at the day of end of RT, 6 weeks and 12 months after end of RT
  The course over time will be described.
Concentration of nitric oxide in the gas phase of the alveolar or acinar region (CANO) | Before start of radiation therapy (RT), at the day of end of RT, 6 weeks and 12 months after end of RT
  The course over time will be described.
Tissue concentration of nitric oxide of the airway wall (CawNO) | Before start of radiation therapy (RT), at the day of end of RT, 6 weeks and 12 months after end of RT
  The course over time will be described.
Airway compartment diffusing capacity of nitric oxide from the of of the airway wall to the gas stream (DawNO) | Before start of radiation therapy (RT), at the day of end of RT, 6 weeks and 12 months after end of RT
  The course over time will be described.
Total flux of nitric oxide in the conducting airway compartment (JawNO) | Before start of radiation therapy (RT), at the day of end of RT, 6 weeks and 12 months after end of RT
  The course over time will be described.
Forced expiratory volume in 1 second | Before start of radiation therapy (RT), at the day of end of RT, 6 weeks and 12 months after end of RT
  The course over time will be described.
Forced vital capacity | Before start of radiation therapy (RT), at the day of end of RT, 6 weeks and 12 months after end of RT
  The course over time will be described.
Forced expiratory flow between 25% and 75% of forced vital capacity | Before start of radiation therapy (RT), at the day of end of RT, 6 weeks and 12 months after end of RT
  The course over time will be described.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No